CLINICAL TRIAL: NCT00267072
Title: The University of Louisville Ovarian Screening Study
Brief Title: Ovarian Screening Study
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 328.01
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives of this study are:

* To identify women at increased risk for developing ovarian cancer
* To detect ovarian cancers at an early stage
* To investigate the role of tumor membrane fragments as tumor markers for early ovarian carcinoma

DETAILED DESCRIPTION:
In the year 2001 approximately 23,400 women in the USA are expected to be diagnosed with ovarian carcinoma and 13,900 will die of the disease. This means that within the USA more women die annually from ovarian cancer than all other gynecologic malignancies combined. Within the Commonwealth of Kentucky approximately 250 women per year develop ovarian carcinoma.

Survival for patients with ovarian cancer is directly related to the stage of disease at diagnosis. Unfortunately, the majority of women present with advanced disease (Stage III and IV) and most of these patients will die of the disease.

The aim of screening for ovarian cancer is to reduce the morbidity and mortality by detecting the disease at an early stage since ovarian cancer detected when disease is confined to the ovary (Stage I) is associated with a dramatically improved 5-year survival. Disease confined to the ovary may be cured in over 90% of patients, in some cases without the need for chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic women over the age of 45 with one or both ovaries.
* Women over the age of 25 with one or both ovaries and any of the following:

  * A personal history of breast, colon or endometrial cancer or breast cancer gene (BRCA) 1 or 2 positive
  * First-degree relative (mother, sister, daughter) with ovarian or breast cancer
  * Two family members with either breast and/or ovarian cancer
  * Mother, sister, daughter, grandparent with a positive BRCA1 or BRCA2 genetic test result.
  * Past use of fertility drugs such as Clomid or Pergonal for more than a year.

Exclusion Criteria:

* Women who are symptomatic of ovarian cancer

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2001-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyril W. Helm, MD, Principal Investigator — University of Louisville, James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Background] Greenlee RT, Hill-Harmon MB, Murray T, Thun M. Cancer statistics, 2001. CA Cancer J Clin. 2001 Jan-Feb;51(1):15-36. doi: 10.3322/canjclin.51.1.15. PMID 11577478